CLINICAL TRIAL: NCT02176642
Title: Double-Blind Randomized Controlled Trial of Extended Release Oxybutynin Versus Placebo in Women Receiving Posterior Tibial Nerve Stimulation for Treatment of Urgency Urinary Incontinence
Brief Title: Comparison of Combination Therapy vs Single Agent Therapy for Treatment of Urge Incontinence.
Acronym: APP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00052742
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Urinary Urge Incontinence
Keywords: Urinary Urge Incontinence; Posterior Tibial Nerve Stimulation; PTNS; Neuromodulation; Oxybutynin; Anticholinergic Medication
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutynin plus PTNS (Active Comparator): Oxybutynin extended release (blinded tablet) 5mg by mouth daily for 6 weeks, Posterior Tibial Nerve Stimulation utilizing the Urgent PC neuromodulation system administered weekly in the office setting for a total of 6 weeks.
  Interventions: Drug: Oxybutynin extended release; Device: Posterior Tibial Nerve Stimulation
- Placebo plus PTNS (Placebo Comparator): Placebo (blinded tablet) taken daily for 6 weeks. Posterior Tibial Nerve Stimulation utilizing the Urgent PC neuromodulation system administered weekly in the office setting for a total of 6 weeks.
  Interventions: Device: Posterior Tibial Nerve Stimulation; Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin extended release — 5mg tablet taken by mouth daily for 6 weeks
  Other Names: Ditropan XL
  Arms: Oxybutynin plus PTNS
Device: Posterior Tibial Nerve Stimulation — In office therapy administered for 30 minutes once every week for a total of 6 weeks
  Other Names: Urgent PC Neuromodulation system
Drug: Placebo — Tablet taken by mouth daily for 6 weeks
  Other Names: Dextrose powder
  Arms: Placebo plus PTNS

SUMMARY:
This is a randomized double-blind placebo-controlled clinical trial of posterior tibial nerve stimulation (PTNS) plus extended release oxybutynin versus PTNS alone (placebo pills) in women undergoing treatment of urgency urinary incontinence (UUI).

The investigators hypothesize that combination therapy with PTNS and anticholinergic medication will result in a significant incremental improvement in UUI symptoms over that achieved with PTNS alone. In addition, the investigators hypothesize that the addition of anticholinergics to PTNS will result in a greater improvement in patients' perception of treatment response, symptom distress, and quality of life than PTNS alone.

Specific Aim 1: To compare the change, from baseline, in mean number of UUI episodes per day using a 3-day bladder diary between PTNS plus anticholinergic medication versus PTNS plus placebo in women undergoing treatment for UUI.

Specific Aim 2: To compare the change, from baseline, in a 24hr pad weight between PTNS plus anticholinergic medication versus PTNS plus placebo.

Specific Aim 3: To compare subjective treatment response, symptoms distress, and quality of life between PTNS plus anticholinergic medication versus PTNS plus placebo utilizing the Patient Global Impression of Improvement (PGI-I) and the Overactive Bladder Questionnaire Short Form (OABq-SF).

An interim analysis will be conducted by an independent entity after 50 participants have completed the study protocol. A Data Safety Monitoring Board is not utilized because the study utilizes FDA approved treatments for urgency urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* > 18 years of age
* > 3 UUI episodes on a 3-day bladder diary
* Urge predominant ( > 50% of total incontinence episodes) urinary incontinence based on a three-day bladder diary
* Existing insurance coverage of PTNS therapy.
* Ability to undergo weekly PTNS treatments in clinic for 6 week period of time and complete all study related items
* Not on an anticholinergic or beta agonist medication or, if they are, willing to undergone a three week washout period prior to randomization

Exclusion Criteria:

* Any previous PTNS therapy, intra-detrusor botulinum toxin injections, or implanted sacral neuromodulation
* Contraindication to anticholinergic therapy (narrow-angle glaucoma or gastric retention) or PTNS therapy (implanted pacemaker/defibrillator or peripheral neuropathy)
* Symptomatic urinary tract infection that has not resolved prior to randomization
* Surgical treatment for stress urinary incontinence or pelvic organ prolapse recommended or planned at time of enrollment
* Surgically altered detrusor muscle
* Known diagnosis or history of neurogenic bladder, post void residual volume >150ml, bladder malignancy, interstitial cystitis/painful bladder syndrome, or pelvic radiation
* Surgery for pelvic organ prolapse or stress urinary incontinence within the previous 3 months
* Pregnancy, lactation, or planned pregnancy during study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazema Y Siddiqui, MD, MHS, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Urogynecology, Durham, North Carolina
  - Duke OB/GYN Consultants of Raleigh, Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified, recruited, and enrolled at the time of their outpatient clinic visits with the Duke Urogynecology clinic. All women who were considering therapy with posterior tibial nerve stimulation were approached for participation in the study.
Pre-assignment Details: A total of 104 patients were assessed for eligibility. Forty-nine patients declined or were deemed ineligible. Fifty-five patients consented to participate but 20 dropped out before randomization. Therefore, a total of 35 patients were randomized as noted in the boxes below (18 in the active medication group, 17 in the placebo group).
Period: Overall Study
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Started | 18 | 17
Completed | 18 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who started treatment were included in analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.8) | 70.4 (8.5) | 71.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Median Number of UUI Episodes Per Day
Description: To compare the change, from baseline, in median number of UUI episodes per day using a 3-day bladder diary between PTNS plus anticholinergic medication versus PTNS plus placebo in women undergoing treatment for UUI. UUI change score will be calculated [post-treatment UUI/day minus pre-treatment UUI/day].
Time Frame: Baseline, 6 weeks
Population: 3 patients in each group did not provide bladder diaries at their 6 week visit, so did not have information available to calculate the primary outcome measure. Median change in UUI episodes/day from baseline to 6 weeks was compared between 2 groups using Wilcoxon Rank Sum test.
Measure: Median (Inter-Quartile Range); unit: Urge urinary incontinence episodes/day
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 15 | 13
Urge urinary incontinence episodes/day | -0.3 [-3.2 to 0.5] | 0.3 [-1 to 1]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Non-Inferiority — We estimated that women in the placebo group would have mean reduction of 3 UUI episodes per day. Assuming 50% improvement in UUI episodes per day is a clinically significant improvement, we estimated the experimental group would have a mean reduction of 4.5 UUI episodes per day with a SD of 1.5 UUI episodes per day. To detect such a difference with 80% power and alpha 0.05, we would need 88 participants for our analysis. To allow for a 12% dropout rate, our goal was to enroll 100 women; p = 0.2, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in 24hr Pad Weight
Description: To compare the change, from baseline, in 24h pad weight between PTNS plus anticholinergic medication versus PTNS plus placebo. Change in median 24h pad weight from baseline to 6 weeks was compared between the 2 groups using Wilcoxon Rank Sum test.
Time Frame: Baseline, 6 weeks
Population: Six participants in the placebo+PNTS group and 3 patients in the oxybutynin+PTNS group did not provide a pad weight at the end of the study, and thus were unable to have the pad weight change score calculated.
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 15 | 10
grams | -52 [-201.5 to -15.1] | -8 [-103.5 to 13.5]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Change in the Patient Global Impression of Improvement (PGI-I)
Description: The Patient Global Impression of Improvement (PGI-I) is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (Very much better to) 7 (Very much worse).
Time Frame: Baseline, 6 weeks
Population: 2 patients in the oxybutynin+PTNS group and one patient in the placebo+PTNS group did not complete the 6 week PGI-I questionnaire so they were not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 16 | 15
units on a scale | -1 [-1 to 0] | -1 [-1 to 0]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Change in the Overactive Bladder Questionnaire Short Form (OABq-SF) Part 1
Description: Part 1 of the OABq-SF questionnaire asks about the relative bother a patient experiences with regard to overactive bladder symptoms over the previous 4 weeks. This part of the questionnaire has 6 questions, with scores ranging from 6 (least amount of bother) to 36 (most amount of bother). For this secondary outcome, we are measuring the change in score on the OABq-SF Part 1 from baseline to 6 weeks. Median change in scores were compared between the 2 groups using Wilcoxon Rank Sum test.
Time Frame: Baseline, 6 weeks
Population: 3 patients in the oxybutynin+PTNS group did not submit their OABq-SF at the end of the study, so they were unable to be included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 15 | 16
units on a scale | -13.3 [-25 to -5.1] | -10 [-23.3 to 6.7]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Change in the Overactive Bladder Questionnaire Short Form (OABq-SF) Part 2
Description: Part 2 of the OABq-SF questionnaire asks about the relative bother a patient experiences with regard to overactive bladder symptoms over the previous 4 weeks. This part of the questionnaire has 13 questions, with scores ranging from 13 (least amount of bother) to 78 (most amount of bother). For this secondary outcome, we are measuring the change in score on the OABq-SF Part 2 from baseline to 6 weeks. Median change in scores were compared between the 2 groups using Wilcoxon Rank Sum test.
Time Frame: Baseline, 6 weeks
Population: Four patients in the oxybutynin+PTNS group and 1 patient in the placebo+PTNS did not submit their OABq-SF part 2 at the end of the study, so they were unable to be included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 14 | 15
units on a scale | 9.2 [6.5 to 18.1] | 0 [-7.7 to 11.6]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Change in the Urinary Distress Inventory (UDI-6)
Description: The UDI-6 is a 6-question inventory of how frequently and how much bother patients have from overactive bladder symptoms. The scores range from 0 (not at all) to 24 (a great deal of bother). We compared the change in scores from baseline to 6 weeks between the 2 groups using Wilcoxon Rank Sum test.
Time Frame: Baseline, 6 weeks
Population: 1 patient in the oxybutynin+PTNS group did not complete the 6 week UDI-6 questionnaire so was not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 17 | 16
units on a scale | -11.1 [-16.6 to 0] | 5.5 [-16.6 to 13.9]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Change in the Incontinence Impact Questionnaire (IIQ-7)
Description: The IIQ-7 is a 7-question score assessing how urinary incontinence affects a patient's various activities and feelings. The range of possible scores is from 0 (not at all) to 28 (a great deal). Median change in scores from baseline to 6 weeks were compared between the 2 groups using Wilcoxon Rank Sum test.
Time Frame: Baseline, 6 weeks
Population: 1 patient in the oxybutynin+PTNS group did not complete the 6 week IIQ-7 questionnaire so was not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 17 | 16
units on a scale | -9.5 [-19 to 0] | -2.4 [-11.9 to 4.8]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Change in Treatment Satisfaction Questionnaire for Medication, Version Two (TSQMvII) - Global Satisfaction Domain
Description: To compare treatment satisfaction between PTNS plus anticholinergic medication versus PTNS plus placebo using the Treatment Satisfaction Questionnaire for Medication, version two (TSQMvII). Patients completed the questionnaire at baseline and again at 6 weeks. The TSQMvII satisfaction domains at each timepjoint were transformed into a score from 0 (extremely dissatisfied) to 100 (extremely satisfied). Median change in scores from baseline to 6 weeks were compared between the 2 groups using Wilcoxon Rank Sum Test.
Time Frame: Baseline, 6 weeks
Population: Two patients in the placebo+PTN group and 1 patient in the oxybutynin+PTNS group did not complete the 6 week TSQMvII questionnaire so was not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 17 | 14
units on a scale | 83.3 [50 to 100] | 70.8 [50 to 83.3]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Change in Treatment Satisfaction Questionnaire for Medication, Version Two (TSQMvII) - Side Effects Domain
Description: To compare bother from medication side effects between PTNS plus anticholinergic medication versus PTNS plus placebo using the Treatment Satisfaction Questionnaire for Medication, version two (TSQMvII). The questionnaire was completed at baseline and at 6 weeks. The TSQMvII side effects domain at each time point was transformed into a score from 0 (extremely dissatisfied) to 150 (extremely satisfied). Median change in scores from baseline to 6 weeks were compared between the 2 groups using Wilcoxon Rank Sum Test.
Time Frame: Baseline, 6 weeks
Population: Two patients in the placebo+PTN group did not complete the 6 week TSQMvII questionnaire so was not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
Number analyzed (Participants) | 18 | 14
units on a scale | 0 [0 to 41.7] | 0 [0 to 50]
Statistical Analysis 1: Comparison: Oxybutynin Plus PTNS vs Placebo Plus PTNS; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline to 6 weeks
Description: We systematically assessed for adverse events related to either PTNS or medication/placebo on a weekly basis. Any adverse events related to PTNS were documented on the patients weekly treatment note for the clinic encounter. Any adverse events related to study medication or placebo were documented via the TSQMvII questionnaire that subjects completed on a weekly basis during treatment.
Arm/Group | Oxybutynin Plus PTNS | Placebo Plus PTNS
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin Plus PTNS (N=18) | Placebo Plus PTNS (N=16)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Possible cardiac symptons (Cardiac disorders) | 0 (0) | 1 (1) — chest pain, shortness of breath, headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes